CLINICAL TRIAL: NCT03710434
Title: A Phase I, Open-Label Study to Assess the Pharmacokinetics and Relative Bioavailability of AZD4635 in Non-Smoking Healthy Male Subjects, With the Option to Assess Food Effect, pH Effect and Absolute Bioavailability
Brief Title: AZD4635 Relative Bioavailability Study
Acronym: Rel Bio
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D8730C00002; 2018-003366-14 (EudraCT Number)
Record Dates: First submitted 2018-10-16; First posted 2018-10-18 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Healthy Volunteers
Keywords: Phase 1, healthy, bioavailability, pharmacokinetics
MeSH Terms: interventions — Lansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Part A - nano-suspension (Experimental): Subjects will receive single dose of AZD4635 50mg nano-suspension (reference) in the fasted state.
  Interventions: Drug: AZD4635 50 mg nano-suspension (reference)
- Part A - solid oral formulation (Experimental): Subjects will receive single dose of AZD4635 50mg solid oral formulation, in the fasted state.
  Interventions: Drug: AZD4635 solid oral formulation - fasted
- Part B-solid oral formulation with food (Experimental): Subjects will receive a single dose AZD4635 solid oral formulation after high fat meal.
  Interventions: Drug: AZD4635 solid oral formulation - fed
- Part B - solid oral formulation with PPI (Experimental): Subjects will receive 30 mg lansoprazole BID and a single dose of AZD4635 solid oral formulation in the fasted state.
  Interventions: Drug: Lansoprazole and AZD4635 50 mg solid oral formulation
- Part B - dose exploration 1 (Experimental): If dose adjustment is required, subjects will receive a different single dose (XX mg) of AZD4635 solid oral formulation, in the fasted state.
  Interventions: Drug: AZD4635 solid oral formulation - fasted
- Part B - dose exploration 2 (Experimental): If dose adjustment is required, subjects will receive a different single dose (YY mg) of AZD4635 solid oral formulation, in the fasted state.
  Interventions: Drug: AZD4635 solid oral formulation - fasted
- Part B - variant 1 (Experimental): Subjects will receive a single dose of AZD4635 solid oral formulation, variant 1 in the fasted state and optional [14C] AZD4635 IV microtracer.
  Interventions: Drug: AZD4635 solid oral formulation variant 1 - fasted; Drug: [14C] AZD4635 IV microtracer - fasted
- Part B - variant 2 (Experimental): Subjects will receive a single dose of AZD4635 solid oral formulation, variant 2 in the fasted state.
  Interventions: Drug: AZD4635 solid oral formulation variant 2 - fasted

INTERVENTIONS:
Drug: AZD4635 50 mg nano-suspension (reference) — Subjects will receive a single dose of AZD4635 50 mg nano-suspension (reference) in the fasted state.
  Arms: Part A - nano-suspension
Drug: AZD4635 solid oral formulation - fasted — Subjects will receive a single dose of AZD4635 solid oral formulation, in the fasted state.
  Arms: Part A - solid oral formulation; Part B - dose exploration 1; Part B - dose exploration 2
Drug: AZD4635 solid oral formulation - fed — Subjects will receive a single dose of AZD4635 solid oral formulation, in the fed state.
  Arms: Part B-solid oral formulation with food
Drug: Lansoprazole and AZD4635 50 mg solid oral formulation — Subjects will receive lansoprazole 30 mg BID for 5 days followed by a single dose of AZD4635 50 mg solid oral formulation in the fasted state.
  Arms: Part B - solid oral formulation with PPI
Drug: AZD4635 solid oral formulation variant 1 - fasted — Subjects will receive a single dose of AZD4635 solid oral formulation, variant 1 in the fasted state.
  Arms: Part B - variant 1
Drug: AZD4635 solid oral formulation variant 2 - fasted — Subjects will receive a single dose of AZD4635 solid oral formulation, variant 2 in the fasted state.
  Arms: Part B - variant 2
Drug: [14C] AZD4635 IV microtracer - fasted — Subjects will receive a single dose of [14C] AZD4635 IV microtracer. This intervention will be co-administered with AZD4635 solid oral formulation variant 1.
  Arms: Part B - variant 1

SUMMARY:
To investigate the pharmacokinetics and relative bioavailability of AZD4635 solid oral formulation and compare with the nano-suspension reference formulation with the option to assess food effect, pH effect and absolute bioavailability

DETAILED DESCRIPTION:
This is a single centre, phase 1, open-label randomised, 2-part study to assess the pharmacokinetics and relative bioavailability of AZD4635 in non-smoking healthy male subjects, with the option to assess food effect, pH effect and absolute bioavailability. It is planned to enrol 20 subjects who will participate in both parts of the study. Subjects will receive a single-dose of AZD4635 in 6 dosing periods with a minimum washout of 9 days between doses.

Part A is a 2-period randomised crossover study of single doses of AZD4635. Subjects will be randomised to receive 50mg AZD4635 nano-suspension (reference) or 50mg AZD4635 solid oral formulation, in the fasted state.

Part B is a 4-period, open-label, randomised, crossover study of single doses of AZD4635 in the same subjects from Part A. The treatments selected for Part B will depend on the outcome of interim analyses of AZD4635 exposure. Subjects will receive 2 of the following 4 treatments in dosing periods 3 and 4:

* A single dose of AZD4635 solid oral formulation dose after a high fat meal
* A single dose of AZD4635 solid oral formulation co-administered with a proton pump inhibitor (PPI), lansoprazole (fasted state)
* A different single dose (XX mg) of AZD4635 solid oral formulation (fasted state)
* Another different single dose (YY mg) of AZD4635 solid oral formulation (fasted state)

Periods 5 and 6 is a 2-period randomised crossover of two variants of AZD4635 solid oral formulation. Subjects will be randomised to receive AZD4635 solid oral formulation variant 1 in the fasted state or AZD4635 solid oral formulation variant 2 in the fasted state. In Periods 5 and 6, Part B an IV microtracer dose of [14C] AZD4635 with solid oral formulation, variant 1 will be administered.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male subjects aged 18 to 55 years with suitable veins for cannulation or repeated venepuncture and IV infusion.
3. Have a body mass index of 18.0 to 32.0 kg/m2, and weigh at least 50 kg and no more than 100 kg.
4. Must be willing and able to communicate and participate in the whole study
5. Must agree to adhere to the contraception requirements, as precaution should avoid fathering a child by either true abstinence or use together, with their female partner/spouse, a highly effective contraception form of birth control in combination with a barrier method, starting from the time of AZD4635 administration until 90 days after the last dose of AZD4635.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which in investigator opinion, may put volunteer at risk because of participation in the study, or influence results of volunteer's ability to participate in the study.
2. History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
3. Presence of refractory nausea and vomiting or chronic gastrointestinal diseases.
4. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
5. Any confirmed clinically significant abnormalities in clinical chemistry, haematology or urinalysis as judged by the investigator
6. Any confirmed clinically significant abnormal findings in vital signs, as judged by investigator.
7. BP >140/90 mmHg or history of hypertension.
8. Any confirmed clinically significant abnormal findings in 12-lead ECG, as judged by investigator.
9. Any positive result at screening for serum hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results.
10. Known or suspected history of drug or alcohol abuse within the past 2 years, as judged by the investigator.
11. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of first administration of IMP in this study. The period of exclusion begins 3 months after the final dose or 1 month after the last visit, whichever is longest. Note: subjects consented and screened, but not randomized in this study or a previous Phase I study are not excluded.
12. Plasma donation within 1 month of screening or any blood donation/loss of more than 500 mL of blood during the 3 months prior to screening.
13. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD4635 or the formulation excipients. Hayfever is allowed unless it is active.
14. Current smokers and those who have smoked within last 12 months. A breath carbon monoxide reading of greater than 10 ppm at screening and admission.
15. Current users of e-cigarettes and nicotine replacement products and those who have used these products within last 12 months.
16. Positive screen for drugs of abuse at screening or admission to the clinical unit or positive screen for alcohol at screening or admission to the clinical unit.
17. Herbal preparations/medications are not allowed throughout the study. These herbal medications include, but are not limited to, St. John's wort, kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone, yohimbe, saw palmetto, and ginseng. Subjects should stop using these herbal medications 14 days prior to the first dose of AZD4635.
18. Use of any prescribed or nonprescribed medication including antacids, H2 antagonists, PPI, analgesics (other than paracetamol/acetaminophen up to 4 g/day), vitamins and minerals during the two weeks prior to first administration of IMP or longer if medication has a longer half-life. Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as agreed by the PI and sponsor's medical monitor.
19. Known or suspected history of alcohol or drug abuse or regular alcohol consumption in males >21 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 Units = 125 mL glass of wine, depending on type)
20. Subjects who are study site employees, or immediate family members of a study site or sponsor employee
21. Subjects who have previously been enrolled in this study or have previously received AZD4635.
22. Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017, shall participate in the study
23. Subjects who have been enrolled in an ADME study in the last 12 months.
24. Subjects with Gilberts Syndrome or a history of cholecystectomy or gall stones.
25. Judgment by investigator that volunteer should not participate in study if they have any ongoing or recent (ie, during the screening period) minor medical complaints that may interfere with the interpretation of the study data or are considered unlikely to comply with the study procedures, restrictions and requirements.
26. Failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 21 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of AZD4635 solid oral formulation and nano-suspension (reference) | Blood samples collected pre-dose, and postdose at 0.25h, 0.5h, 1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h, 96h and 120h
  Assessment of maximum concentration (Cmax) in plasma
Exposure to AZD4635 solid oral formulation and nano-suspension (reference) | Blood samples collected pre-dose, and postdose at 0.25h, 0.5h, 1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h, 96h and 120h
  Assessment of exposure through measurement of area under the curve (AUC) in plasma

SECONDARY OUTCOMES:
Time to maximum concentration (tmax) of AZD4635 solid oral formulation variants 1 and 2 in plasma | Blood samples collected pre-dose, and postdose at 0.25h, 0.5h, 1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h, 96h and 120h
  Assessment of time to maximum concentration (tmax) in plasma
Maximum concentration (Cmax) of AZD4635 solid oral formulation variants 1 and 2 in plasma | Blood samples collected pre-dose, and postdose at 0.25h, 0.5h, 1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h, 96h and 120h
  Assessment of maximum concentration (Cmax) in plasma
Area under the plasma concentration-time curve from zero to time of last measurable concentration (AUClast) for AZD4635 solid oral formulation variants 1 and 2 | Blood samples collected pre-dose, and postdose at 0.25h, 0.5h, 1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h, 96h and 120h
  Assessment of exposure through measurement of area under the curve (AUClast) in plasma
Area under the plasma concentration-time curve from zero to 48 hours (AUC 0-48) for AZD4635 solid oral formulation variants 1 and 2 | Blood samples collected pre-dose, and postdose at 0.25h, 0.5h, 1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h and 48h
  Assessment of exposure through measurement of area under the curve (AUC 0-48) in plasma
Area under the plasma concentration-time curve from zero to infinity (AUC 0-inf.) for AZD4635 solid oral formulation variants 1 and 2 | Blood samples collected pre-dose, and postdose at 0.25h, 0.5h, 1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h, 96h and 120h
  Exposure to AZD4635 through measurement of area under the curve (AUC 0-inf.) in plasma
Determine absolute bioavailability (F) of AZD4635 | Predose, 0.25h, 0.33h, 0.42h, 0.5h, 0.58h, 0.67h, 0.75h, 1h, 1.25h, 1.5h, 2h, 2.5h, 4.5h, 6.5h, 8.5h, 12.5h, 24h 48h, 72h, 96h, 120h
  Absolute bioavailability (F) will be calculated from area under the plasma concentration versus time curve (AUC) of the oral dose of AZD4635/ AUC of the IV dose of [14C]AZD4635 x IV dose/oral dose /100
Time to maximum concentration (tmax) of AZD4635 solid oral formulation in plasma in fasted and fed state (optional) | Blood samples collected pre-dose, and postdose at 0.25h, 0.5h, 1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h, 96h and 120h
  Assessment of time to maximum concentration (tmax) in plasma in fasted and fed state
Maximum concentration (Cmax) of AZD4635 solid oral formulation in plasma in fasted and fed state (optional) | Blood samples collected pre-dose, and postdose at 0.25h, 0.5h, 1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h, 96h and 120h
  Assessment of maximum concentration (Cmax) in plasma in fasted and fed state
Area under the plasma concentration-time curve from zero to time of last measurable concentration (AUClast) for AZD4635 solid oral formulation in fasted and fed state (optional) | Blood samples collected pre-dose, and postdose at 0.25h, 0.5h, 1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h, 96h and 120h
  Assessment of exposure in fasted and fed state through measurement of area under the curve (AUClast) in plasma
Area under the plasma concentration-time curve from zero to 48 hours (AUC 0-48) for AZD4635 solid oral formulation in fasted and fed state (optional) | Blood samples collected pre-dose, and postdose at 0.25h, 0.5h, 1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h and 48h
  Assessment of exposure in fasted and fed state through measurement of area under the curve (AUC 0-48) in plasma
Area under the plasma concentration-time curve from zero to infinity (AUC 0-inf.) for AZD4635 solid oral formulation in fasted and fed state (optional) | Blood samples collected pre-dose, and postdose at 0.25h, 0.5h, 1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h, 96h and 120h
  Assessment of exposure in fasted and fed state through measurement of area under the curve (AUC 0-inf.) in plasma
Time to maximum concentration (tmax) of AZD4635 solid oral formulation with and without lansoprazole PPI (proton pump inhibitor) (optional) | Blood samples collected pre-dose, and postdose at 0.25h, 0.5h, 1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h, 96h and 120h
  Assessment of time to maximum concentration (tmax) in plasma
Maximum concentration (Cmax) of AZD4635 solid oral formulation with and without lansoprazole PPI (proton pump inhibitor) (optional) | Blood samples collected pre-dose, and postdose at 0.25h, 0.5h, 1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h, 96h and 120h
  Assessment of maximum concentration (Cmax) in plasma
Area under the plasma concentration-time curve from zero to time of last measurable concentration (AUClast) for AZD4635 solid oral formulation with and without lansoprazole PPI (proton pump inhibitor) (optional) | Blood samples collected pre-dose, and postdose at 0.25h, 0.5h, 1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h, 96h and 120h
  Assessment of exposure through measurement of area under the curve (AUClast) in plasma
Area under the plasma concentration-time curve from zero to 48 hours (AUC 0-48) for AZD4635 solid oral formulation with and without lansoprazole PPI (proton pump inhibitor) (optional) | Blood samples collected pre-dose, and postdose at 0.25h, 0.5h, 1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h and 48h
  Assessment of exposure through measurement of area under the curve (AUC 0-48) in plasma
Area under the plasma concentration-time curve from zero to infinity (AUC 0-inf.) for AZD4635 solid oral formulation with and without lansoprazole PPI (proton pump inhibitor) (optional) | Blood samples collected pre-dose, and postdose at 0.25h, 0.5h, 1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h, 96h and 120h
  Assessment of exposure through measurement of area under the curve (AUC 0-inf.) in plasma
Number of adverse events (AE) experienced by subjects | Approximately 6 months
  Safety and tolerability assessed through incidence of AE

CONTACTS AND LOCATIONS:
Overall Officials: Sharan Sidhu, MBChB, BAO, MRCS, MFPM, Principal Investigator — Quotient Sciences Limited (indemnified by Medical Protection Society)
Locations (1):
- Research Site, Ruddington, United Kingdom

REFERENCES:
- See also: Results of this clinical trial are available on www.astrazenecaclinicaltrials.com — https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Search